CLINICAL TRIAL: NCT06368453
Title: A Study to Evaluate the Performance, Usability, and Result Interpretation of INSTI® HIV Self-Test When Performed by Observed Intended Users in the US
Brief Title: A Study to Evaluate the Performance, Usability, and Result Interpretation of INSTI® HIV Self-Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: bioLytical Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: CLS-003
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Human Immunodeficiency Virus I Infection; Human Immunodeficiency Virus II Infection
Keywords: HIV Self Test; INSTI HIV Self test; HIV-1/2 Antibody Test; In-Home HIV test

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Performance (Experimental): INSTI® HIV ST devices are provided to the enrolled participants to conduct the self test using the provided instruction for use while being observed by an operator. The operator records the INSTI® HIV ST results interpreted by the subjects. The operator then performs the comparator test to compare the results with the INSTI® HIV ST.
  Interventions: Device: INSTI® HIV Self-Test
- Mock results interpretation study and Usability evaluation (No Intervention): A subset of the enrolled subjects (500 subjects) will participate in the mock results interpretation study and usability evaluation. For the mock study, the subjects will be presented with 5 mock INSTI® HIV ST devices with different results, and the subject's interpretation of each device will be recorded. The percentage of subjects who interpreted the mock results correctly for each result type will be calculated.
  For the INSTI® HIV ST usability evaluation, the subjects will be presented with a questionnaire. The overall results of the questionnaire will be used to determine the percentage of subjects who found the INSTI® HIV ST easy to use.

INTERVENTIONS:
Device: INSTI® HIV Self-Test — Each participant will be provided with the INSTI® HIV Self-Test and asked to conduct self testing. The operator will observe the participant and record the subject's interpretation of the results. Subjects will perform the test without intervention from the operator.
  The operator will then perform the comparator test and collect a fingerstick blood sample. In the event of a discrepant result between the INSTI® HIV ST and comparator test, an additional venous blood sample will be collected from the subject and sent for discrepancy testing.
  Arms: Performance

SUMMARY:
The objective of this study is to evaluate the performance, usability, and result interpretation of the INSTI® HIV Self-Test (referred to INSTI® HIV ST) in the intended use population across the United States (US). The INSTI® HIV Self-Test is a single use in vitro test that is used as a self-test for the detection of antibodies to HIV-1 and HIV-2 in human fingerstick blood. This study is designed to evaluate INSTI® HIV ST performance in the hands of non-professionals and untrained lay users who are inexperienced in HIV blood-based self-testing.

The study aims to:

To evaluate the clinical performance (i.e., diagnostic sensitivity and specificity) of the INSTI® HIV Self-Test in a lay user population.

To assess the user's comprehension of the INSTI® HIV ST results (e.g., interpreting positive, negative, and invalid results).

To evaluate the usability of the INSTI® HIV ST and understand users' experience in performing the test.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the performance, usability, and result interpretation of the INSTI® HIV Self-Test (referred to INSTI® HIV ST) in the intended user population across the United States (US). This study is designed to evaluate INSTI® HIV ST performance in the hands of non-professionals and untrained lay users who are inexperienced in HIV self-testing.

The study aims to:

To evaluate the clinical performance (i.e., diagnostic sensitivity and specificity) of the INSTI® HIV ST in a lay user population.

To assess the user's comprehension of the INSTI® HIV ST results (e.g., interpreting positive, negative, and invalid results).

To evaluate the usability of the INSTI® HIV ST and understand users' experience in performing the test.

Subjects will be consecutively enrolled from the 'general' population (i.e., "all comers" group of previously undiagnosed HIV individuals) until a minimum of 27 HIV positive and 1000-1700 HIV negatives are obtained. Subjects will be lay users recruited at multiple sites across the US. This study is to determine if lay users, unassisted, can perform the INSTI® HIV ST correctly and without significant risk of incorrect results. The study will help to determine if the INSTI® HIV ST instructions are easy to understand for the US public. The overall study processes include a performance evaluation, where subjects will perform the INSTI® HIV ST, a mock results interpretation study to assess the user's comprehension of the INSTI® HIV ST results and usability evaluation to understand users experience with the INSTI® HIV ST. Only a subset of the enrolled subjects (500 subjects) will participate in the mock results interpretation study and usability evaluation.

For the performance evaluation, subjects will perform the INSTI® HIV ST without any intervention from an observer. Following the subjects self-testing, an operator will collect an additional fingerstick sample to perform a comparator test. The positive and negative percent agreement (i.e., PPA and NPA) between the INSTI® HIV ST result and comparator will be calculated. In the event of discrepant results between the INSTI® HIV ST and comparator test, an additional venous blood sample will be collected from the subject for discrepancy testing.

A subset of the enrolled subjects will then participate in the mock results interpretation study and usability evaluation. For the mock study, the subjects will be presented with 5 mock INSTI® HIV ST devices with different results, and the subject's interpretation of each device will be recorded. The percentage of subjects who interpreted the mock results correctly for each result type will be calculated.

For the INSTI® HIV ST usability evaluation, the subjects will be presented with a questionnaire. The overall results of the questionnaire will be used to determine the percentage of subjects who found the INSTI® HIV ST easy to use.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Operator/study staff must complete the subject's Enrolment Questionnaire
* Subject to sign and date the Informed Consent Form
* Able to complete the required testing on the allocated testing day(s).
* Able to speak/ read/write English or Spanish
* Willingness to provide the fingerstick blood sample and if necessary, the volume of whole blood collected through venous blood draw (approximately 7 ml)
* Willingness to participate in the study site's standard of care HIV counselling and testing program and receive the study site's standard of care test results
* Unknown HIV Status

Exclusion Criteria:

* Has participated in any prior, or concurrent trial of HIV self-tests
* Is a practicing medical healthcare professional (doctor, nurse or HIV Counsellor that performs HIV testing with Rapid Tests)
* Is currently on a PrEP regimen
* Has used a Rapid Diagnostic Test for HIV blood-based self-testing previously
* Has received any experimental HIV vaccine
* Has a bleeding disorder
* Is known HIV+
* Uses Anti-Retroviral medication
* Any condition which, in the opinion of the Operator, would make the participant unsuitable or unsafe for enrolment or could interfere with the completion of the assessment, consent form and questionnaire etc. or bias the outcome, i.e., being unable to see / read by forgetting to bring reading glasses, being intoxicated or acute sickness, or visibly distressed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1728 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2025-01-08 (Actual); Study Completion 2025-01-08 (Actual)

PRIMARY OUTCOMES:
Clinical sensitivity and specificity of the INSTI® HIV Self-Test | 12 Months
  The positive percent agreement (PPA) and negative percent agreement (NPA) between the INSTI® HIV ST and comparator test will be determined. The two-sided confidence interval for the PPA and NPA will be determined.
  The percentage of assays with INSTI® HIV ST invalid results will be determined.

SECONDARY OUTCOMES:
The INSTI® HIV Self-Test usability and result interpretation | 12 Months
  The percentage of subjects who interpreted the INSTI® HIV ST mock results correctly for each result type will be determined.
  The usability questionnaire will be used to determine the following:
  The percentage of subjects who found the INSTI® HIV ST easy to use. The percentage of subjects who found the INSTI® HIV ST product information easy to use.
  The percentage of subjects willing to use the INSTI® HIV ST again The percentage of subjects willing to recommend the INSTI® HIV ST

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Geller, Principal Investigator — Centennial Medical Group; Anthony LaMarca, Principal Investigator — Therafirst Medical Centers Inc.
Locations (1):
- Therafirst Medical Center, Fort Lauderdale, Florida, United States